CLINICAL TRIAL: NCT06091878
Title: Gene Expression Profiling in a Validation Cohort of Locally Advanced and Recurrent/Metastatic Salivary Gland Cancers: The INDAGA-UK Trial
Brief Title: Gene Expression Profiling in a Validation Cohort of Locally Advanced and Recurrent/Metastatic Salivary Gland Cancers
Acronym: INDAGA-UK
Status: Not yet recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5899
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Salivary Gland Cancer
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observational study, no intervention

SUMMARY:
The INDAGA-UK trial is a retrospective, multi-centre observational study in participants with locally advanced and recurrent salivary gland to investigate t its molecular profiling, and to explore new prognostic and druggable markers. We will analyse samples and data from patients diagnosed with salivary gland cancer from 2013 - 2023. Subject and sample identification will occur over a 12-month period. Samples and data will be analysed over the next 12 months prior to study end.

ELIGIBILITY:
Inclusion Criteria:

1. Aged over 18
2. Histological diagnosis of salivary gland cancer (SGCs)
3. Availability of archival tissue (acceptable after 2013 up to present)
4. Ability to give informed consent (if applicable)* for retrieving histological specimen and preform molecular analysis *De-identified archival tissue from deceased patients will be collected as part of the study once REC approval is in place, if the patient was alive when the samples were taken and they are not part of the NHS opt out scheme.

Exclusion Criteria:

1. Different H&N cancer of other histology
2. Thyroid cancers

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants with a salivary gland cancer diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
• Description of the molecular and genomic profile of locally advanced and recurrent-metastatic SGCs. | Time Frame: Through study completion, expected duration of 10 years
  • Description of the molecular and genomic profile of locally advanced and recurrent-metastatic SGCs.

IPD SHARING:
Plan to Share IPD: Undecided